CLINICAL TRIAL: NCT02905136
Title: Mechanisms of Auto-immune Encephalitis
Acronym: MECANO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0439
Record Dates: First submitted 2016-07-04; First posted 2016-09-19 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Autoimmune Encephalitis
Keywords: autoantibodies; neuronal synaptic receptors; autoimmune encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, whole blood, cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with confirmed diagnosis of autoimmune encephalitis by: Patient with confirmed diagnosis of autoimmune encephalitis by French rare disease reference center on PNS with :
  * with detection in CSF of characterized antibodies against neuronal synaptic receptor or protein (anti-NMDAr, anti-LGI1, anti-CASPR2, Anti-AMPAr, anti-mGluR5, anti-GABAbr)
  * or uncharacterized antibodies
  Interventions: Other: Fundamental research

INTERVENTIONS:
Other: Fundamental research — serum, whole blood, cerebrospinal fluid

SUMMARY:
Neurological and psychiatric diseases are one of the major health problems worldwide. Decades of fundamental and clinical research have led to the model that these disorders results from synaptic imbalance between excitatory, inhibitory and modulatory systems in key brain structures. Although the network and neurotransmitter systems involved have been delineated, the mechanisms leading to improper neurotransmissions remain poorly understood. One major limitation lays in the difficulty to transpose the identified dysregulation in humans to relevant animal models in which molecular and cellular targets can be manipulated.

The amino-acid glutamate mediates the vast majority of excitatory neurotransmission in the mammalian brain. We know that the glutamatergic synapses can change their strength by regulating surface expression and dynamics of their postsynaptic receptors, through changes in receptor recycling and/or lateral diffusion. This synaptic plasticity underlies higher cognitive functions such as learning and memory and is likely compromised in several disease states. Regulating glutamate receptor number and function is thus of primary importance. New subcellular imaging technique rendered possible the study of receptor trafficking and receptor regulation in various conditions including pathological models opening new fundamental questions. Moreover, recent breakthroughs on glutamate receptor structure offer unprecedented clues on the molecular and structural mechanisms underpinning receptor dysfunction at the atomic level.

Recently, description of encephalitis associated with specific autoantibodies (Abs) directed against neuronal synaptic receptors or proteins (NSA-Abs) opens new lights in the pathophysiological mechanisms of some human brain disorders. The best example and the most frequent syndrome is the synaptic autoimmune encephalitis associated with autoantibodies against extracellular domains of the glutamatergic NMDA receptor (NMDAR-Abs). Classically, patients first present psychiatric symptoms with hallucinations and bizarre behavior before development of neurological symptoms such as seizures, dyskinesia, and autonomic instability. Despite the severity of neuropsychiatric symptoms, more than 80% of patients fully recover after immunomodulatory treatments and many arguments suggest a direct role of NMDAR-Abs in the symptoms. The investigators recently demonstrated that NMDAR-Abs directly modify, at the synaptic level, NMDAR lateral diffusion by disruption of the interaction between NMDAR and EphrinB2 receptor, a synaptic protein anchoring NMDAR at the synapse (Mikasova et al, Brain 2012; Dupuis et al, EMBOJ 2014). These data suggest that NMDAR-Abs could directly participate in the neuropsychiatric disorders observed in patients and that NMDAR dysfunctions could be directly responsible for the observed symptoms. Furthermore, these data suggest that other NSA-Abs directed against other synaptic proteins could explain specific neurological symptoms in patients with encephalitis that are not associated with NMDAR-Abs.

The aim of MECANO is to combine multidisciplinary approaches (clinical, immunological, and neurobiological ones) to identify new NSA-Abs, to characterize their specific pathological roles and to decipher acute and chronic NMDAR-Abs effects on biophysical and structural properties of the NMDA receptor, synaptic plasticity, neuronal morphology, and cognitive performance. This project should provide key insights onto the effects of patients' NSA-Abs on the cellular dynamic and regulation of synaptic proteins or receptors and on the molecular cascades activated during synapse dysfunction. The investigators will investigate how NSA-Abs binding alter receptor activity, modify surface receptor mobility and dynamically regulate the maturation of synapses and circuitries. For that purpose, The investigators will use a unique combination of high-resolution imaging (single nanoparticle tracking), receptor engineering, cellular electrophysiology, computational (structural modeling) and cellular and molecular biology approaches and finally behaviour assays. Based on both cutting-edge neurobiology and clinical expertise of autoimmune disorders, and strengthened by promising preliminary experiments, the MECANO project will likely open new avenues of fundamental research in the understanding of synaptic dysfunction and clinical research for the treatment of neuropsychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* No age limit
* Diagnosis of autoimmune encephalitis with detection in CSF of characterized antibodies against neuronal synaptic receptor or uncharacterized antibodies
* Written inform consent form
* Affiliated to social security institution
* Availability of surplus biological samples (serum and CSF)

Exclusion Criteria:

* Other cause of encephalitis (infectious, toxic, metabolic, vascular)
* Impairment of surplus biological samples
* Refusal by the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with confirmed diagnosis of autoimmune encephalitis by French rare disease reference center on PNS with :
  * with detection in CSF of characterized antibodies against neuronal synaptic receptor or protein (anti-NMDAr, anti-LGI1, anti-CASPR2, Anti-AMPAr, anti-mGluR5, anti-GABAbr)
  * or uncharacterized antibodies
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Pathophysiological study of interaction between specific autoantibodies neuronal synaptic receptors in autoimmune encephalitis : in vivo model | through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Honnorat, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Institut NeuroMyoGène Équipe Synaptopathies et Autoanticorps (SynatAc) INSERM U1217 / UMR CNRS 5310, Bron, France